CLINICAL TRIAL: NCT04212286
Title: A Single-Center, Prospective Study Comparing the Diagnostic Efficiencies of Contrast-Enhanced Ultrasound and EOB Contrast-Enhanced Magnetic Resonance Imaging for Lesions With Diameters ≤ 2cm in Patients With High Risk of HCC
Brief Title: Comparing the Diagnostic Efficiencies of CEUS and EOB-MRI in Patients With High Risk of HCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Third Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: drjingxiang002
Record Dates: First submitted 2019-12-02; First posted 2019-12-26 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Hepatocellular Cancer; Liver Cirrhoses; Diagnoses Disease
Keywords: Hepatocellular Cancer; Contrast-enhanced ultrasound; EOB-MRI; Diagnostic Efficacy
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic CEUS and EOB-MRI (Experimental): Patients with high risk of HCC having suspicious lesions with Diameters ≤ 2cm will receive CEUS and EOB-MRI examinations.
  Interventions: Diagnostic Test: Diagnostic CEUS and EOB-MRI

INTERVENTIONS:
Diagnostic Test: Diagnostic CEUS and EOB-MRI — Undergo Sonovue-CEUS and EOB-MRI

SUMMARY:
HCC is a serious threat to the health of people. Accurate diagnosis of early HCC by imaging allows patients to obtain proper treatment. However, for lesions with diameters ≤2 cm, the tumor blood supply is not fully established, and there may be no typical manifestation on the image. In addition, atypical enhanced patterns caused by liver cirrhosis may also hinder imaging diagnosis of HCC. Therefore, early diagnosis of HCC in the context of cirrhosis remains a major clinical problem.

Contrast-enhanced Ultrasound (CEUS) and MRI Contrast-enhanced Magnetic Resonance Imaging (CEMRI) are common diagnostic imaging methods. Till now, there is still lack of a detailed investigation comparing the diagnostic efficacies of CEUS and EOB-MRI for micro HCC in the context of cirrhosis. Therefore, this study aims to analyze the imaging patterns in CEUS and EOB-MRI for liver lesions with diameters ≤ 2 cm among patients with high risk of HCC, and to compare the diagnostic efficacies of EOB-MRI and CEUS for early-stage HCCs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are at high risk of HCC.
2. The ages of patients are between 18 and 80.
3. Patients are with solid liver lesion(s) ≤ 2 cm detected by imaging scan (US/CT/MRI).
4. The number of lesions is less than or equal to 3.
5. Patient is able and willing to receive CEUS and EOB-MRI examinations within 30 days.
6. Patient signs the informed consent.

Exclusion Criteria:

1. Patient is with lesions confirmed by pathology or follow-up, or hemangiomas.
2. Patient is with lesions already undergoing local treatment, including thermal ablation or TACE.
3. Patient is with severe cardiopulmonary insufficiency.
4. Patient is a pregnant or breastfeeding women.
5. Patient is considered to be unsuitable to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
The sensitivity, specificity and accuracy of CEUS and EOB-MRI | 6 to 12 months
  The sensitivity, specificity and accuracy of CEUS and EOB-MRI for liver lesion ≤ 2 cm will be calculated.

SECONDARY OUTCOMES:
The sensitivity, specificity and accuracy of combined CEUS and EOB-MRI | 6 to 12 months
  The sensitivity, specificity and accuracy of combined CEUS and EOB-MRI for liver lesion ≤ 2 cm will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Jing, MD, Study Director — Tianjin Third Central Hospital
Locations (1):
- Tianjin Third Central Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qin Z, Zhou Y, Zhang X, Ding J, Zhou H, Wang Y, Zhao L, Chen C, Jing X. The comparison of contrast-enhanced ultrasound and gadoxetate disodium-enhanced MRI LI-RADS for nodules </=2 cm in patients at high risk for HCC: a prospective study. Front Oncol. 2024 May 7;14:1345981. doi: 10.3389/fonc.2024.1345981. eCollection 2024. PMID 38774417